CLINICAL TRIAL: NCT00367939
Title: An Multicenter Study to Evaluate the Efficacy and Safety of a 5 Week Therapy With the Combination of Valsartan 160 mg Plus Amlodipine 10 mg in Hypertensive Patients Not Adequately Responding to a 5 Week Therapy With Ramipril 5 mg and Felodipine 5 mg
Brief Title: Efficacy and Safety of the Combination of Valsartan Plus Amlodipine in Hypertensive Patients Not Adequately Responding to the Combination Therapy With Ramipril Plus Felodipine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVAA489ADE01
Record Dates: First submitted 2006-08-22; First posted 2006-08-24 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine, Valsartan Drug Combination

INTERVENTIONS:
Drug: valsartan + amlodipine

SUMMARY:
The purpose of this study is to evaluate the efficacy of valsartan plus amlodipine in hypertensive patients not responding to treatment with ACE inhibitor plus calcium channel blocker

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients (18 years or older)
* Females must be either post-menopausal for one year, surgically sterile or using effective contraceptive methods (e.g. barrier method with spermicide, intra-uterine device, hormonal contraceptives).
* Patients with moderate essential hypertension (WHO II)

Exclusion Criteria:

* Severe hypertension
* Pregnant or nursing women
* Treated hypertensive patients with controlled hypertension under current therapy (MSDBP < 90 mmHg and MSSBP < 140 mmHg)
* A history of cardiovascular disease, including angina pectoris, myocardial infarction, coronary artery bypass graft, percutaneous transluminal coronary angioplasty, transient ischemic attack, stroke, and heart failure NYHA II - IV
* Other protocol-defined exclusion criteria may apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2005-12; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
To investigate whether 5 weeks of treatment with valsartan 160mg + amlodipine 10mg provide add'l mean sitting systolic BP reduction in patients not adequately responding to 5 weeks of treatment with ramipril + felodipine--i.e., mean systolic BP

SECONDARY OUTCOMES:
To evaluate the effects of valsartan 160 mg plus amlodipine 10 mg on mean sitting diastolic BP, normalization and responder rate.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma Ag, Study Director — Novartis Pharmaceuticals
Locations (1):
- Investigative Centers, Germany

REFERENCES:
- [Derived] Trenkwalder P, Schaetzl R, Borbas E, Handrock R, Klebs S. Combination of amlodipine 10 mg and valsartan 160 mg lowers blood pressure in patients with hypertension not controlled by an ACE inhibitor/CCB combination. Blood Press Suppl. 2008 Dec;2:13-21. doi: 10.1080/08038020802488855. PMID 19205092